CLINICAL TRIAL: NCT04335318
Title: Real Life AI in Polyp Detection
Acronym: RELIANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Alexander Hann, Principal Investigator, Wuerzburg University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AI01
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Colonic Polyp
Keywords: Deep Learning; Polyp detection rate; CNN
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colonoscopy with AI-assistance group (Experimental): Colonoscopies were performed with AI-assistance.
  Interventions: Device: AI-assisted colonoscopy
- Standard Colonoscopy group (No Intervention): Standard clinical procedure

INTERVENTIONS:
Device: AI-assisted colonoscopy — Colonoscopies performed with assistance of an AI tool that highlights the areas that are susceptible to be a polyp.
  Arms: Colonoscopy with AI-assistance group

SUMMARY:
The objective of this study is to compare the polyp detection rate (PDR) of endoscopists unaware of a commercially available artificial intelligence (AI) device for polyp detection during colonoscopy and the PDR of endoscopists with the aid of such a device. Moreover, an extensive characterization of the performance of this device will be done.

DETAILED DESCRIPTION:
Recently, there have been remarkable breakthroughs in the introduction of deep learning techniques, especially convolutional neural networks (CNNs), in assisting clinical diagnosis in different medical fields. One of these artificial intelligence (AI) devices to diagnose colon polyps during colonoscopy was launched in October 2019. Its intended use is to work as an adjunct to the endoscopist during a colonoscopy with the purpose of highlighting regions with visual characteristics consistent with different types of mucosal abnormalities.

It is essential to know whether deep learning algorithms can really help endoscopists during colonoscopies. Several studies have already addressed this issue with different approaches and results. However, one common drawback of these type of Machine vs Human retrospective studies is endoscopist bias. It is usually generated because of human natural competitive spirit against machine or human relaxation because of AI-reliance. This can have an effect in the overall results.

The investigators perfomed colonoscopies with the use of a commercially available AI system to detect colonic polyps and recorded them during clinical routine. Additionally from March 2019 - May 2019, 120 colonoscopy videos were performed and captured prospectively without the use of AI.

In this study, the investigators plan to retrospectively compare those two video sets regarding the polyp detection rate, withdrawal time and polyp identification characteristics of the AI system.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopies for Polyp detection

Exclusion Criteria:

* Colonoscopies for Inflammatory Bowel Disease (IBD).
* Colonoscopies for work up of an active bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Polyp detection rate comparison | 45 minutes
  Number of polyps detected divided by number of colonoscopies
Mean withdrawal time comparison | 45 minutes
  Mean withdrawal time comparison

SECONDARY OUTCOMES:
AI-Polyp bounding boxes - True Positive Evaluation | 45 minutes
  2 approaches: frame by frame analysis and temporal coherence analysis
AI-Polyp bounding boxes - False Positive Quantitative Evaluation | 45 minutes
  3 approaches depending on window-time detection
AI-Polyp bounding boxes - False Negative Evaluation | 45 minutes
  Number of by bounding box missed polyps
Reaction Time Analysis | 45 minutes
  Comparison time of polyp detection in a human vs machine approach

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hann, PD Dr. Med, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- Universitätsklinikum Würzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No